CLINICAL TRIAL: NCT02943629
Title: A "Less-rapid" Sequence Anesthetic Induction/Intubation Sequence? Does Apneic Oxygenation by Means of an Oxygenating Laryngoscope Blade Prolong the "Duration of Apnea Without Desaturation" in Paralyzed Non-obese and Morbidly Obese Patients?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of feasibility
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Curtis Baysinger, Professor of Anesthesiology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160579
Record Dates: First submitted 2016-10-20; First posted 2016-10-25 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Apneic Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Non-Obese: Apneic Oxygenation: eight minute (Experimental): Non-obese healthy female patients requiring endotracheal anesthesia for gynecologic (open or laparoscopic) abdominal surgery will have the Pentax AWSTM video laryngoscope with attached P blade placed and then receive 10 l/minute flow of oxygen through the P blade (apneic oxygenation) for eight minutes, or earlier if SpO2 falls to ≤ 95%. The trachea will then be intubated and the ventilation of the lungs will commence using 100% oxygen until SpO2 ≥ 98%.
  Interventions: Device: Apneic oxygenation: Eight minute
- Non-Obese: Without Apneic Oxygenation (Other): Non-obese healthy female patients requiring endotracheal anesthesia for gynecologic (open or laparoscopic) abdominal surgery will have the Pentax AWSTM video laryngoscope with attached P blade placed for eight minutes, or earlier if SpO2 falls to ≤ 95%. The trachea will then be intubated and the ventilation of the lungs will commence using 100% oxygen until SpO2 ≥ 98%.
  Interventions: Device: Without apneic oxygenation
- Obese: Apneic Oxygenation: five minute (Experimental): Morbidly obese patients (BM I ≥ 40 kg/m2) requiring endotracheal anesthesia for gynecologic (open or laparoscopic) abdominal surgery will have the Pentax AWSTM video laryngoscope with attached P blade placed and then receive 10 l/minute flow of oxygen through the P blade (apneic oxygenation) for five minutes, or earlier if SpO2 falls to ≤ 95%. The trachea will then be intubated and the ventilation of the lungs will commence using 100% oxygen until SpO2 ≥ 98%.
  Interventions: Device: Apneic oxygenation: five minutes
- Obese: Without Apneic Oxygenation (Other): Morbidly obese patients (BM I ≥ 40 kg/m2) requiring endotracheal anesthesia for gynecologic (open or laparoscopic) abdominal surgery will have the Pentax AWSTM video laryngoscope with attached P blade placed for five minutes, or earlier if SpO2 falls to ≤ 95%. The trachea will then be intubated and the ventilation of the lungs will commence using 100% oxygen until SpO2 ≥ 98%.
  Interventions: Device: Without apneic oxygenation

INTERVENTIONS:
Device: Apneic oxygenation: Eight minute — A Pentax AWSTM video laryngoscope with attached P blade will be placed and then 10 l/minute flow of oxygen will be administered through the P blade (apneic oxygenation) for eight minutes, or less if SpO2 falls to ≤ 95%. The trachea will then be intubated and the ventilation of the lungs will commence using 100% oxygen until SpO2 ≥ 98%.
  Arms: Non-Obese: Apneic Oxygenation: eight minute
Device: Without apneic oxygenation — A Pentax AWSTM video laryngoscope with attached P blade will be placed for eight minutes, or less if SpO2 falls to ≤ 95%. The trachea will then be intubated and the ventilation of the lungs will commence using 100% oxygen until SpO2 ≥ 98%.
  Arms: Non-Obese: Without Apneic Oxygenation; Obese: Without Apneic Oxygenation
Device: Apneic oxygenation: five minutes — A Pentax AWSTM video laryngoscope with attached P blade will be placed and then 10 l/minute flow of oxygen will be administered through the P blade (apneic oxygenation) for five minutes, or less if SpO2 falls to ≤ 95%. The trachea will then be intubated and the ventilation of the lungs will commence using 100% oxygen until SpO2 ≥ 98%.
  Arms: Obese: Apneic Oxygenation: five minute

SUMMARY:
The study will test the efficacy of the Pentax AWSTM video laryngoscope (VLS) equipped with a P Blade (Figure 1) as the means to provide Apneic Oxygenation (AO) and prolong Duration of Apnea Without Desaturation (DAWD) in non-obese and morbidly obese females.

DETAILED DESCRIPTION:
Pre-oxygenation/de-nitrogenation for three minutes of spontaneous breathing or alternatively four to eight deep breaths prior to rapid sequence anesthetic induction/intubation (RSII) in patients with healthy lungs, low oxygen demands and normal hemoglobin levels allows up to eight minutes of safe apnea time or DAWD.

The study will test the efficacy of the Pentax AWSTM video laryngoscope (VLS) equipped with a P Blade as the means to provide apneic oxygenation and prolong DAWD. The P Blade sports a suction conduit which can equally well provide a conduit for oxygen administration. The initial phase of the study will include non-obese healthy (ASAR 1-2) women patients requiring endotracheal anesthesia for gynecologic (open or laparoscopic) abdominal surgery. Subsequently a cohort of morbidly obese patients (BM I ≥ 40 kg/m2) also requiring gynecologic abdominal access will be recruited for investigation.

Participants of each group (obese, non-obese) will be randomized to apneic oxygenation with the the Pentax AWS Laryngoscope or no apneic oxygenation.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients,
2. American Society of Anesthesiologists Rating 1-2,
3. Aged 18 through 65 years of age
4. Elective gynecological surgery via an abdominal approach (laparoscopic or open)
5. Already consented to general anesthesia necessitating endotracheal intubation.
6. Are candidates for anesthesia using laryngeal mask airway if needed

Exclusion Criteria:

1. Patient refusal to enter study
2. History of difficult mask ventilation
3. History of, or anticipated difficult intubation
4. Heavy Smokers (> 10 cigarettes per day)
5. Asthma
6. Chronic Obstructive Pulmonary Disease
7. Heart Disease
8. Renal or Liver disease
9. Neurological disease.
10. Women scored at ≥ 3/4 on the modified Mallampati scale 30.
11. Women exhibiting other signs of a potential difficult intubation (limited neck flexion or extension; neck circumference > 30 cm; prominent incisors)
12. Patients with a baseline resting oxygenation level of less than 95%.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Duration of apnea without desaturation | Time in seconds from the initiation of laryngoscopy until the time at which Sp02 falls to 95%, or until 8 minutes have elapsed

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Baysinger, MD, Principal Investigator — Vanderbilt University Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] FRUMIN MJ, EPSTEIN RM, COHEN G. Apneic oxygenation in man. Anesthesiology. 1959 Nov-Dec;20:789-98. doi: 10.1097/00000542-195911000-00007. No abstract available. PMID 13825447
- [Background] Paolini JB, Donati F, Drolet P. Review article: video-laryngoscopy: another tool for difficult intubation or a new paradigm in airway management? Can J Anaesth. 2013 Feb;60(2):184-91. doi: 10.1007/s12630-012-9859-5. Epub 2012 Dec 12. PMID 23233395
- [Background] Tanoubi I, Drolet P, Donati F. Optimizing preoxygenation in adults. Can J Anaesth. 2009 Jun;56(6):449-66. doi: 10.1007/s12630-009-9084-z. Epub 2009 Apr 28. PMID 19399574
- [Background] Jense HG, Dubin SA, Silverstein PI, O'Leary-Escolas U. Effect of obesity on safe duration of apnea in anesthetized humans. Anesth Analg. 1991 Jan;72(1):89-93. doi: 10.1213/00000539-199101000-00016. PMID 1984382
- [Background] Shah U, Wong J, Wong DT, Chung F. Preoxygenation and intraoperative ventilation strategies in obese patients: a comprehensive review. Curr Opin Anaesthesiol. 2016 Feb;29(1):109-18. doi: 10.1097/ACO.0000000000000267. PMID 26545146
- [Background] Weingart SD, Levitan RM. Preoxygenation and prevention of desaturation during emergency airway management. Ann Emerg Med. 2012 Mar;59(3):165-75.e1. doi: 10.1016/j.annemergmed.2011.10.002. Epub 2011 Nov 3. PMID 22050948
- [Background] De Jong A, Molinari N, Pouzeratte Y, Verzilli D, Chanques G, Jung B, Futier E, Perrigault PF, Colson P, Capdevila X, Jaber S. Difficult intubation in obese patients: incidence, risk factors, and complications in the operating theatre and in intensive care units. Br J Anaesth. 2015 Feb;114(2):297-306. doi: 10.1093/bja/aeu373. Epub 2014 Nov 27. PMID 25431308
- [Background] Gebremedhn EG, Mesele D, Aemero D, Alemu E. The incidence of oxygen desaturation during rapid sequence induction and intubation. World J Emerg Med. 2014;5(4):279-85. doi: 10.5847/wjem.j.issn.1920-8642.2014.04.007. PMID 25548602
- [Background] Altermatt FR, Munoz HR, Delfino AE, Cortinez LI. Pre-oxygenation in the obese patient: effects of position on tolerance to apnoea. Br J Anaesth. 2005 Nov;95(5):706-9. doi: 10.1093/bja/aei231. Epub 2005 Sep 2. PMID 16143575
- [Background] Archer GW Jr, Marx GF. Arterial oxygen tension during apnoea in parturient women. Br J Anaesth. 1974 May;46(5):358-60. doi: 10.1093/bja/46.5.358. No abstract available. PMID 4157184
- [Background] McClelland SH, Bogod DG, Hardman JG. Apnoea in pregnancy: an investigation using physiological modelling. Anaesthesia. 2008 Mar;63(3):264-9. doi: 10.1111/j.1365-2044.2007.05347.x. PMID 18289232
- [Background] McClelland SH, Bogod DG, Hardman JG. Pre-oxygenation and apnoea in pregnancy: changes during labour and with obstetric morbidity in a computational simulation. Anaesthesia. 2009 Apr;64(4):371-7. doi: 10.1111/j.1365-2044.2008.05785.x. PMID 19317700
- [Background] Patil S, Sinha P, Krishnan S. Successful delivery in a morbidly obese patient after failed intubation and regional technique. Br J Anaesth. 2007 Dec;99(6):919-20. doi: 10.1093/bja/aem326. No abstract available. PMID 18006534
- [Background] Hawkins JL, Chang J, Palmer SK, Gibbs CP, Callaghan WM. Anesthesia-related maternal mortality in the United States: 1979-2002. Obstet Gynecol. 2011 Jan;117(1):69-74. doi: 10.1097/AOG.0b013e31820093a9. PMID 21173646
- [Background] Teller LE, Alexander CM, Frumin MJ, Gross JB. Pharyngeal insufflation of oxygen prevents arterial desaturation during apnea. Anesthesiology. 1988 Dec;69(6):980-2. doi: 10.1097/00000542-198812000-00035. No abstract available. PMID 3195773
- [Background] Ramachandran SK, Cosnowski A, Shanks A, Turner CR. Apneic oxygenation during prolonged laryngoscopy in obese patients: a randomized, controlled trial of nasal oxygen administration. J Clin Anesth. 2010 May;22(3):164-8. doi: 10.1016/j.jclinane.2009.05.006. PMID 20400000
- [Background] Baraka AS, Taha SK, Siddik-Sayyid SM, Kanazi GE, El-Khatib MF, Dagher CM, Chehade JM, Abdallah FW, Hajj RE. Supplementation of pre-oxygenation in morbidly obese patients using nasopharyngeal oxygen insufflation. Anaesthesia. 2007 Aug;62(8):769-73. doi: 10.1111/j.1365-2044.2007.05104.x. PMID 17635423
- [Background] El-Orbany M, Connolly LA. Rapid sequence induction and intubation: current controversy. Anesth Analg. 2010 May 1;110(5):1318-25. doi: 10.1213/ANE.0b013e3181d5ae47. Epub 2010 Mar 17. PMID 20237045
- [Background] Hayes AH, Breslin DS, Mirakhur RK, Reid JE, O'Hare RA. Frequency of haemoglobin desaturation with the use of succinylcholine during rapid sequence induction of anaesthesia. Acta Anaesthesiol Scand. 2001 Jul;45(6):746-9. doi: 10.1034/j.1399-6576.2001.045006746.x. PMID 11421834
- [Background] Taha SK, El-Khatib MF, Baraka AS, Haidar YA, Abdallah FW, Zbeidy RA, Siddik-Sayyid SM. Effect of suxamethonium vs rocuronium on onset of oxygen desaturation during apnoea following rapid sequence induction. Anaesthesia. 2010 Apr;65(4):358-61. doi: 10.1111/j.1365-2044.2010.06243.x. PMID 20402874
- [Background] Tang L, Li S, Huang S, Ma H, Wang Z. Desaturation following rapid sequence induction using succinylcholine vs. rocuronium in overweight patients. Acta Anaesthesiol Scand. 2011 Feb;55(2):203-8. doi: 10.1111/j.1399-6576.2010.02365.x. PMID 21226862
- [Background] Achar SK, Pai AJ, Shenoy UK. Apneic Oxygenation during simulated prolonged difficult laryngoscopy: Comparison of nasal prongs versus nasopharyngeal catheter: A prospective randomized controlled study. Anesth Essays Res. 2014 Jan-Apr;8(1):63-7. doi: 10.4103/0259-1162.128911. PMID 25886106
- [Background] Wimalasena Y, Burns B, Reid C, Ware S, Habig K. Apneic oxygenation was associated with decreased desaturation rates during rapid sequence intubation by an Australian helicopter emergency medicine service. Ann Emerg Med. 2015 Apr;65(4):371-6. doi: 10.1016/j.annemergmed.2014.11.014. Epub 2014 Dec 20. PMID 25536868
- [Background] Patel A, Nouraei SA. Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE): a physiological method of increasing apnoea time in patients with difficult airways. Anaesthesia. 2015 Mar;70(3):323-9. doi: 10.1111/anae.12923. Epub 2014 Nov 10. PMID 25388828
- [Background] Harbut P, Gozdzik W, Stjernfalt E, Marsk R, Hesselvik JF. Continuous positive airway pressure/pressure support pre-oxygenation of morbidly obese patients. Acta Anaesthesiol Scand. 2014 Jul;58(6):675-80. doi: 10.1111/aas.12317. Epub 2014 Apr 16. PMID 24738713
- [Background] Mitterlechner T, Herff H, Hammel CW, Braun P, Paal P, Wenzel V, Benzer A. A dual-use laryngoscope to facilitate apneic oxygenation. J Emerg Med. 2015 Jan;48(1):103-7. doi: 10.1016/j.jemermed.2014.06.061. Epub 2014 Oct 11. PMID 25308899
- [Background] Yentis SM, Lee DJ. Evaluation of an improved scoring system for the grading of direct laryngoscopy. Anaesthesia. 1998 Nov;53(11):1041-4. doi: 10.1046/j.1365-2044.1998.00605.x. PMID 10023271
- [Background] Samsoon GL, Young JR. Difficult tracheal intubation: a retrospective study. Anaesthesia. 1987 May;42(5):487-90. doi: 10.1111/j.1365-2044.1987.tb04039.x. PMID 3592174